CLINICAL TRIAL: NCT03457207
Title: Combined Mini Laparotomy With Laparoscopy Appraoch for Management of Endometrioma
Brief Title: Mini Laparotomy With Laparoscopy for Management of Endometrioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30
Record Dates: First submitted 2018-02-25; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined minilaparotomy- laparoscopy approach (Experimental): women undergo the new technique of surgical treatment of endometriomas of the ovary
  Interventions: Procedure: Combined minilaparotomy- laparoscopy approach

INTERVENTIONS:
Procedure: Combined minilaparotomy- laparoscopy approach — Laparoscopic aspiration of cyst then guided its extracorporeal cystectomy then reposition and evaluation by laproscopy

SUMMARY:
Under general anaesthesia, the patient is placed in the modified dorsal lithotomy position a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).

Aspiration of the cyst:

Veress needle is inserted in the midline 2 cm above the symphysis pubis to aspirate the cyst under laparoscopic guidance (to guide the entry of the needle into the cyst wall & to confirm complete aspiration).

Delivery of affected ovary outside the abdominal cavity:

Classic ovarian cystectomy will be done using microsurgical techniques in which the cyst wall will be dissected gently and carefully from the healthy ovarian tissue followed by perfect haemostasis and re-fashioning of the remaining ovarian tissue using Vicryl (3-0) sutures.

Re-introduction of the ovary to inside the abdominal cavity:

The stitched ovary is pushed gently inside the abdominal cavity and the minilaparotomy is re-covered by the rubber shield (to allow re-inflation of the abdominal cavity). The ovary is reassessed under laparoscopic guidance to ensure perfect haemostasis and normal position of the ovary. Pelvic irrigation is done if needed.

DETAILED DESCRIPTION:
Under general anaesthesia, the patient is placed in themodified dorsal lithotomy position (to ensure lax anterior abdominal wall). The patient is thenprepped and draped in the usual fashion for an abdominaland vaginal procedure. In non- virgin patients, vaginal speculum is inserted into thevagina to expose the cervix, a uterine manipulator is inserted in the cervix followed by placement of a Foley's catheter in thebladder. As regards port placement, a 10-mm umbilical trocar is inserted. A panoramic view of the pelvis was obtained together with full assessment of the ovarian mass(es).

Aspiration of the cyst:

Veress needle is inserted in the midline 2 cm above the symphysis pubis to aspirate the cyst under laparoscopic guidance (to guide the entry of the needle into the cyst wall & to confirm complete aspiration).

Delivery of affected ovary outside the abdominal cavity:

A transverse mini-laparotomy is done (2-3 cm) in the midline 2 cm above the symphysis pubis. A long shanks artery forceps is introduced inside the abdominal cavity (to grasp the affected ovary) under laparoscopic guidance. Then, the artery is pulled gently to the outside to deliver the ovary at the minilaparotomy skin incision. Careful handling and traction is applied to avoid injury of both the ovarian tissue or/andinfundibulopelvic ligament. Following the delivery of the ovary, the abdominal incision is temporary closed using (Eshaped 10 x 10 cm) rubbershield (to avoid any soiling of abdominal cavity with blood or cystic fluid & give the chance to reinflate the abdominal cavity later on).

Ovarian cystectomy:

Classic ovarian cystectomy will be done using microsurgical techniques in which the cyst wall will be dissected gently and carefully from the healthy ovarian tissue followed by perfect haemostasis and re-fashioning of the remaining ovarian tissue using Vicryl (3-0) sutures.The stitched ovary is pushed gently inside the abdominal cavity and the minilaparotomy is re-covered by the rubber shield (to allow re-inflation of the abdominal cavity). The ovary is reassessed under laparoscopic guidance to ensure perfect haemostasis and normal position of the ovary. Pelvic irrigation is done if needed

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral ovarian endometriotic cysts (≥ 10 cm),
* recurrent ovarian cysts
* good ovarian reserve (antimullerian hormone {AMH} > 1 ng/ml & antral follicular count {AFC} > 4)

Exclusion Criteria:

* solid ovarian masses
* patients who were unfit for surgery
* chronic diseases (e.g. cardiac disease or diabetes)
* any contraindication for laparoscopic surgery (excessive anterior abdominal wall scarring)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2015-01-02 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Recurrance | 2 years after surgery
  reappearance of endometriomas in the ipsilateral ovary

SECONDARY OUTCOMES:
Ovarian reserve | 6 months after surgery
  Measurment of day 2 serum FSH
Ovarian reserve | 6 months after surgery
  measurment of AMH
ovarian reserve | 6 months after surgery
  Measurement of antral follicular count

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided